CLINICAL TRIAL: NCT04020419
Title: Natural Berry Extract Treatment of Hemangiomas
Acronym: Pediaberry
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study ending early due to program transferring to another site.
Sponsor: Gayle Gordillo (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Gayle Gordillo, Professor, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1810087420; 2R01GM095657 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-07-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hemangioma
Keywords: miR126; Pediaberry
MeSH Terms: conditions — Hemangioma

STUDY DESIGN:
Intervention Model Description: pilot study to determine effect size for possible FDA phase I/II trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: investigational pharmacy will have access to randomization schemes and will package study drug from bulk supplies. All other study team members and participants are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pediaberry group (Experimental): PediaBerry™ is a proprietary blend powdered berry extracts
  Interventions: Drug: PediaBerry
- Placebo (Placebo Comparator): Placebo: powdered sugar plus McCormick Color from Nature Food Colors Berry and Sky Blue powdered food color (https://www.mccormick.com/spices-and-flavors/extracts-and-food-colors/food-colors/color-from-nature-assorted-food-color ).
  Interventions: Drug: PediaBerry

INTERVENTIONS:
Drug: PediaBerry — PediaBerry or placebo will be mixed with a cream vehicle for topical administration or with water for oral administration
  Other Names: placebo

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled parallel group study evaluating the use of PediaBerry for the treatment of hemangiomas in infants ≤ 4 months of corrected gestation age over a 6-month treatment period. Subjects will be followed to age 18 months. A total of 44 subjects will be PediaBerry group and 22 subjects in the placebo control group.

DETAILED DESCRIPTION:
PediaBerry™ is a proprietary blend of powdered berry extracts. Placebo: powdered sugar plus McCormick Color from Nature Food Colors Berry and Sky Blue powdered food color (https://www.mccormick.com/spices-and-flavors/extracts-and-food-colors/food-colors/color-from-nature-assorted-food-color ).

Cream vehicle is mixed with PediaBerry™ or placebo at the time of application.Children will receive once daily topical and oral gavage dosing of PediaBerry or placebo.

The first study visit will take place within 2 weeks of subject recruitment. The subject enrollment, consenting and randomization will occur as study visit #0 and will occur at Riley Children's Hospital or Nationwide Children's Hospital. Data collection will be the same at all study visits starting with study visit #1 until the completion of the study. The first dose of PediaBerry™ or placebo will be administered prior to completion of study visit #1, and will also be given at study visits #2-6. Study visits #2-6 will occur monthly study visits until the subject completes 6 months of treatment.Subjects will be weighed and treatment doses adjusted accordingly. Study visits #7-11 to watch for signs of rebound hemangioma proliferation will occur every other month until age 12 months and then at age 15 and 18 months. Urine samples, photos and caliper measurements will occur at each study visit. Some subjects may have less than 11 study visits depending on the age at the time of subject enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Children with hemangiomas ≤ 4 months and 2 weeks of corrected gestational age
* Hemangioma size ≥ 1 cm diameter

Exclusion Criteria:

* Children with hemangiomas that threaten the life of the child or development of vital structures.
* Children who are breast feeding and mother is taking beta blocker medication
* Children with previously treated hemangiomas
* Congenital hemangiomas - cannot distinguish between rapidly involuting and non-involuting congenital hemangiomas
* Hemangiomas located in the perineal/diapering area - product will get contaminated or wiped off with diapering
* Children with food allergies to blueberries or any other kind of berry
* Legal guardian unable to provide informed consent

Ages: 1 Month to 19 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Decreased Hemangioma Size | 6 month treatment period
  Decrease in the size of hemangioma > 50%

SECONDARY OUTCOMES:
Decreased urinary micro RNA 126 levels | 6 month treatment period
  Urinary micro RNA 126 levels are analyzed using quantitative polymerase chain reactions

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Gordillo, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Riley Hospital for Children, Indianapolis, Indiana
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoak JC, Warner ED, Cheng HF, Fry GL, Hankenson RR. Hemangioma with thrombocytopenia and microangiopathic anemia (Kasabach-Merritt syndrome): an animal model. J Lab Clin Med. 1971 Jun;77(6):941-50. No abstract available. PMID 5105323
- [Background] Gordillo G, Fang H, Khanna S, Harper J, Phillips G, Sen CK. Oral administration of blueberry inhibits angiogenic tumor growth and enhances survival of mice with endothelial cell neoplasm. Antioxid Redox Signal. 2009 Jan;11(1):47-58. doi: 10.1089/ars.2008.2150. PMID 18817478
- [Background] Gordillo G, Fang H, Park H, Roy S. Nox-4-dependent nuclear H2O2 drives DNA oxidation resulting in 8-OHdG as urinary biomarker and hemangioendothelioma formation. Antioxid Redox Signal. 2010 Apr 15;12(8):933-43. doi: 10.1089/ars.2009.2917. PMID 19817625
- [Background] Gordillo GM, Atalay M, Roy S, Sen CK. Hemangioma model for in vivo angiogenesis: inducible oxidative stress and MCP-1 expression in EOMA cells. Methods Enzymol. 2002;352:422-32. doi: 10.1016/s0076-6879(02)52038-3. No abstract available. PMID 12125369
- [Background] Gordillo GM, Biswas A, Khanna S, Pan X, Sinha M, Roy S, Sen CK. Dicer knockdown inhibits endothelial cell tumor growth via microRNA 21a-3p targeting of Nox-4. J Biol Chem. 2014 Mar 28;289(13):9027-38. doi: 10.1074/jbc.M113.519264. Epub 2014 Feb 4. PMID 24497637
- [Background] Gordillo GM, Onat D, Stockinger M, Roy S, Atalay M, Beck FM, Sen CK. A key angiogenic role of monocyte chemoattractant protein-1 in hemangioendothelioma proliferation. Am J Physiol Cell Physiol. 2004 Oct;287(4):C866-73. doi: 10.1152/ajpcell.00238.2003. Epub 2004 May 26. PMID 15163622
- [Background] Biswas A, Khanna S, Roy S, Pan X, Sen CK, Gordillo GM. Endothelial cell tumor growth is Ape/ref-1 dependent. Am J Physiol Cell Physiol. 2015 Sep 1;309(5):C296-307. doi: 10.1152/ajpcell.00022.2015. Epub 2015 Jun 24. PMID 26108661
- [Background] Biswas A, Pan X, Meyer M, Khanna S, Roy S, Pearson G, Kirschner R, Witman P, Faith EF, Sen CK, Gordillo GM. Urinary Excretion of MicroRNA-126 Is a Biomarker for Hemangioma Proliferation. Plast Reconstr Surg. 2017 Jun;139(6):1277e-1284e. doi: 10.1097/PRS.0000000000003349. PMID 28538565
- [Background] Atalay M, Gordillo G, Roy S, Rovin B, Bagchi D, Bagchi M, Sen CK. Anti-angiogenic property of edible berry in a model of hemangioma. FEBS Lett. 2003 Jun 5;544(1-3):252-7. doi: 10.1016/s0014-5793(03)00509-x. PMID 12782326
- [Background] Biswas A, Clark EC, Sen CK, Gordillo GM. Phytochemical Inhibition of Multidrug Resistance Protein-1 as a Therapeutic Strategy for Hemangioendothelioma. Antioxid Redox Signal. 2017 Jun 10;26(17):1009-1019. doi: 10.1089/ars.2016.6881. Epub 2016 Nov 9. PMID 27706944
- [Background] Gordillo GM, Biswas A, Khanna S, Spieldenner JM, Pan X, Sen CK. Multidrug Resistance-associated Protein-1 (MRP-1)-dependent Glutathione Disulfide (GSSG) Efflux as a Critical Survival Factor for Oxidant-enriched Tumorigenic Endothelial Cells. J Biol Chem. 2016 May 6;291(19):10089-103. doi: 10.1074/jbc.M115.688879. Epub 2016 Mar 9. PMID 26961872
- [Background] Bruckner AL, Frieden IJ. Hemangiomas of infancy. J Am Acad Dermatol. 2003 Apr;48(4):477-93; quiz 494-6. doi: 10.1067/mjd.2003.200. PMID 12664009
- [Background] Dinehart SM, Kincannon J, Geronemus R. Hemangiomas: evaluation and treatment. Dermatol Surg. 2001 May;27(5):475-85. doi: 10.1046/j.1524-4725.2001.00227.x. PMID 11359498
- [Background] Drolet BA, Esterly NB, Frieden IJ. Hemangiomas in children. N Engl J Med. 1999 Jul 15;341(3):173-81. doi: 10.1056/NEJM199907153410307. No abstract available. PMID 10403856
- [Background] Metry DW, Hebert AA. Benign cutaneous vascular tumors of infancy: when to worry, what to do. Arch Dermatol. 2000 Jul;136(7):905-14. doi: 10.1001/archderm.136.7.905. PMID 10890993
- [Background] Chiller KG, Passaro D, Frieden IJ. Hemangiomas of infancy: clinical characteristics, morphologic subtypes, and their relationship to race, ethnicity, and sex. Arch Dermatol. 2002 Dec;138(12):1567-76. doi: 10.1001/archderm.138.12.1567. PMID 12472344
- [Background] Bauman NM, McCarter RJ, Guzzetta PC, Shin JJ, Oh AK, Preciado DA, He J, Greene EA, Puttgen KB. Propranolol vs prednisolone for symptomatic proliferating infantile hemangiomas: a randomized clinical trial. JAMA Otolaryngol Head Neck Surg. 2014 Apr;140(4):323-30. doi: 10.1001/jamaoto.2013.6723. PMID 24526257
- [Background] Tozzi A. Oral Propranolol for Infantile Hemangioma. N Engl J Med. 2015 Jul 16;373(3):284. doi: 10.1056/NEJMc1503811. No abstract available. PMID 26176393
- [Background] Leaute-Labreze C, Hoeger P, Mazereeuw-Hautier J, Guibaud L, Baselga E, Posiunas G, Phillips RJ, Caceres H, Lopez Gutierrez JC, Ballona R, Friedlander SF, Powell J, Perek D, Metz B, Barbarot S, Maruani A, Szalai ZZ, Krol A, Boccara O, Foelster-Holst R, Febrer Bosch MI, Su J, Buckova H, Torrelo A, Cambazard F, Grantzow R, Wargon O, Wyrzykowski D, Roessler J, Bernabeu-Wittel J, Valencia AM, Przewratil P, Glick S, Pope E, Birchall N, Benjamin L, Mancini AJ, Vabres P, Souteyrand P, Frieden IJ, Berul CI, Mehta CR, Prey S, Boralevi F, Morgan CC, Heritier S, Delarue A, Voisard JJ. A randomized, controlled trial of oral propranolol in infantile hemangioma. N Engl J Med. 2015 Feb 19;372(8):735-46. doi: 10.1056/NEJMoa1404710. PMID 25693013
- [Background] Langley A, Pope E. Propranolol and central nervous system function: potential implications for paediatric patients with infantile haemangiomas. Br J Dermatol. 2015 Jan;172(1):13-23. doi: 10.1111/bjd.13379. Epub 2014 Dec 10. PMID 25175684
- [Background] Barlow CF, Priebe CJ, Mulliken JB, Barnes PD, Mac Donald D, Folkman J, Ezekowitz RA. Spastic diplegia as a complication of interferon Alfa-2a treatment of hemangiomas of infancy. J Pediatr. 1998 Mar;132(3 Pt 1):527-30. doi: 10.1016/s0022-3476(98)70034-4. PMID 9544915
- [Background] Marczylo TH, Cooke D, Brown K, Steward WP, Gescher AJ. Pharmacokinetics and metabolism of the putative cancer chemopreventive agent cyanidin-3-glucoside in mice. Cancer Chemother Pharmacol. 2009 Nov;64(6):1261-8. doi: 10.1007/s00280-009-0996-7. Epub 2009 Apr 11. PMID 19363608
- [Background] Fang J. Bioavailability of anthocyanins. Drug Metab Rev. 2014 Nov;46(4):508-20. doi: 10.3109/03602532.2014.978080. Epub 2014 Oct 27. PMID 25347327
- [Background] Manach C, Williamson G, Morand C, Scalbert A, Remesy C. Bioavailability and bioefficacy of polyphenols in humans. I. Review of 97 bioavailability studies. Am J Clin Nutr. 2005 Jan;81(1 Suppl):230S-242S. doi: 10.1093/ajcn/81.1.230S. PMID 15640486
- [Background] Mahmood I. Application of allometric principles for the prediction of pharmacokinetics in human and veterinary drug development. Adv Drug Deliv Rev. 2007 Sep 30;59(11):1177-92. doi: 10.1016/j.addr.2007.05.015. Epub 2007 Aug 16. PMID 17826864
- [Background] Sharma V, McNeill JH. To scale or not to scale: the principles of dose extrapolation. Br J Pharmacol. 2009 Jul;157(6):907-21. doi: 10.1111/j.1476-5381.2009.00267.x. Epub 2009 Jun 5. PMID 19508398
- [Background] Chang LC, Haggstrom AN, Drolet BA, Baselga E, Chamlin SL, Garzon MC, Horii KA, Lucky AW, Mancini AJ, Metry DW, Nopper AJ, Frieden IJ; Hemangioma Investigator Group. Growth characteristics of infantile hemangiomas: implications for management. Pediatrics. 2008 Aug;122(2):360-7. doi: 10.1542/peds.2007-2767. PMID 18676554
- [Background] Garzon MC, Drolet BA, Baselga E, Chamlin SL, Haggstrom AN, Horii K, Lucky AW, Mancini AJ, Metry DW, Newell B, Nopper AJ, Frieden IJ; Hemangioma Investigator Group. Comparison of infantile hemangiomas in preterm and term infants: a prospective study. Arch Dermatol. 2008 Sep;144(9):1231-2. doi: 10.1001/archderm.144.9.1231. No abstract available. PMID 18794478

DOCUMENTS (1):
  • Informed Consent Form (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT04020419/ICF_000.pdf